CLINICAL TRIAL: NCT03116893
Title: Effect of P-gp Inhibition, OATP-inhibition and Food on the Kinetics of a Single Oral Dose BI 685509 in Healthy Male Subjects
Brief Title: Drug-drug Interaction (DDI) With a P-gp Inhibitor, Organic Anion Transporting Polypeptide OATP-inhibitor, Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1366-0010; 2016-003310-27 (EudraCT Number)
Record Dates: First submitted 2017-04-06; First posted 2017-04-17 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Reference Treatment (Experimental): BI 685509 given alone, fasted
  Interventions: Drug: BI 685509 Fasted Conditions
- Treatment 1 (Experimental): BI 685509, given alone, after a high fat, high calorie breakfast
  Interventions: Drug: BI 685509 After Standardised Breakfast
- Treatment 2 (Experimental): BI 685509, given together with itraconazole, fasted
  Interventions: Drug: Itraconazole
- Treatment 3 (Experimental): BI 685509, given together with rifampicin, fasted
  Interventions: Drug: Rifampin

INTERVENTIONS:
Drug: BI 685509 After Standardised Breakfast — High-fat high calorie breakfast
  Arms: Treatment 1
Drug: Itraconazole — Administration of itraconazole together with BI 685509
  Arms: Treatment 2
Drug: Rifampin — Administration of rifampicin together with BI 685509
  Arms: Treatment 3
Drug: BI 685509 Fasted Conditions — BI 685509, given alone
  Arms: Reference Treatment

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailability of BI 685509 given alone under fasted conditions (Reference, R) compared to the intake after a high fat, high caloric breakfast (Test 1, T1), to combined administration with itraconazole under fasted conditions (Test 2, T2) and to combined administration with rifampin under fasted conditions (Test 3, T3).

The secondary objective is the evaluation and comparison of several pharmacokinetic parameters between the treatments.

DETAILED DESCRIPTION:
BI 685509 is a substrate of the drug transporters P-gp and Organic anion transporting polypeptide 1B1 and 1B3 (OATP1B1/OATP1B3). Inhibition of these transport proteins may result in an increased drug exposure which might impact the safety of the patients. Therefore this trial should investigate whether and to what extent the inhibition of P-gp (mediated by itraconazole) and the inhibition of OATP1B1/OATP1B3 (mediated by rifampin) affects kinetics of BI 685509. Itraconazole and rifampin are recommended probe drugs to test in-vivo inhibition of P-gp and OATP1B1/OATP1B3.

Furthermore the food effect will be investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigators assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure [BP], Pulse Rate [PR]), 12 lead Electrocardiogram [ECG], and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* Body Mass Index [BMI] of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice [GCP] and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure [BP], Pulse Rate [PR] or Electrocardiogram [ECG]) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 60 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. Time between start of the Q-wave and the end of the T-wave in an electrocardiogram/ corrected QT interval [QT/QTc] interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 24 g per day for males)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or any other relevant Electrocardiogram [ECG] finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | 4 Days
  AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)
Cmax (maximum measured concentration of the analyte in plasma) | 4 Days
  Cmax (maximum measured concentration of the analyte in plasma)

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | 4 Days
  AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No